CLINICAL TRIAL: NCT03328533
Title: Norepinephrine Versus Phenylephrine Continuous Variable Infusion for Prevention of Post-spinal Hypotension During Cesarean Delivery: A Randomized Controlled Double-blinded Trial
Brief Title: Norepinephrine Versus Phenylephrine Continuous Variable Infusion in Cesarean Delivery
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Ahmed Hasanin, Assistant professor, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: N-82-2017
Record Dates: First submitted 2017-10-30; First posted 2017-11-01 (Actual); Last update posted 2018-07-17 (Actual); Status verified 2018-07

CONDITIONS: Cesarean Section Complications; Spinal Anesthesia
MeSH Terms: interventions — Phenylephrine; Norepinephrine; Bupivacaine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Phenylephrine (Active Comparator): Will receive spinal anesthesia using Bupivacaine. Then, phenylephrine infusion by a starting rate of 0.75 mcg/Kg/min. The rate will be then adjusted according to the patient blood pressure. The infusion will stop in case of reactive hypertension. The infusion will start again when blood pressure returns to normal reading. Infusion will be increased by 20% if hypotension occurred.
  Interventions: Drug: Phenylephrine; Drug: Bupivacaine
- Norepinephrine (Experimental): Will receive spinal anesthesia using Bupivacaine. Then, norepinephrine bitartrate infusion by a starting rate of 0.1 mcg/Kg/min (equivalent to norepinephrine base of 0.05 mcg/Kg/min). The rate will be then adjusted according to the patient blood pressure. The infusion will stop in case of reactive hypertension. The infusion will start again when blood pressure returns to normal reading. Infusion will be increased by 20% if hypotension occurred.
  Interventions: Drug: Norepinephrine; Drug: Bupivacaine

INTERVENTIONS:
Drug: Phenylephrine — Phenylephrine variable infusion with a starting rate of 0.75 mcg/Kg/min.
  Arms: Phenylephrine
Drug: Norepinephrine — Norepinephrine bitartrate variable infusion with a starting rate of 0.1 mcg/Kg/min (equivalent to norepinephrine base of 0.05 mcg/Kg/min).
  Other Names: Levophed
  Arms: Norepinephrine
Drug: Bupivacaine — Bupivacaine will be injected in the subarachnoid space with a dose of 10 mg.
  Other Names: Marcaine

SUMMARY:
Comparison will be conducted between continuous variable infusions of Phenylephrine with starting dose of 0.75 mcg/Kg/min and Norepinephrine Bitartrate with starting dose of 0.1 mcg/Kg/min (with norepinephrine base of 0.05 mcg/Kg/min) for prophylaxis against Post-spinal hypotension during cesarean delivery

DETAILED DESCRIPTION:
Maternal hypotension is a common complication after spinal anesthesia for cesarean delivery (CD). Many vasopressors have been used for prevention of post-spinal hypotension (PSH) during CD; however, the optimum protocol for prophylaxis is not established yet. Phenylephrine (PE) is a popular vasopressor used in obstetric anesthesia; however, its use is limited by its marked cardiac depressant nature. Norepinephrine (NE) is a potent vasopressor characterized by both α adrenergic agonistic activity in addition to a weak β adrenergic agonistic activity; thus, NE is considered a vasopressor with minimal cardiac depressant effect; these pharmacological properties would make NE an attractive alternative to PE. In this study, the investigators will compare continuous variable infusion of both drugs (PE and NE) with doses of 0.75 mcg/Kg/min and 0.05 mcg/Kg/min respectively for prophylaxis against PSH during CD. We used Norepinephrine Bitartrate 8 mg ampules which contains norepinephrine base of 4 mg.

ELIGIBILITY:
Inclusion Criteria:

* Full term
* Pregnant women
* Scheduled for cesarean section

Exclusion Criteria:

* Pre-eclampsia
* Eclampsia
* Bleeding
* Cardiac dysfunction

Ages: 18 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 123 (Actual)
Dates: Start 2017-11-10 (Actual); Primary Completion 2018-05-01 (Actual); Study Completion 2018-05-05 (Actual)

PRIMARY OUTCOMES:
Incidence of post-spinal anesthesia hypotension. | 30 minutes after spinal anesthesia
  Defined as the percentage of patients with decreased systolic blood pressure less than 80% of the baseline reading

SECONDARY OUTCOMES:
Incidence of severe post-spinal anesthesia hypotension | 30 minutes after spinal anesthesia
  Defined as the percentage of patients with decreased systolic blood pressure less than 60% of the baseline reading
Incidence of severe delivery hypotension | 10 minutes after delivery
  Defined as the percentage of patients with decreased systolic blood pressure less than 80% of the baseline reading
Systolic blood pressure | 2 hours after subarachnoid block
  Systolic blood pressure measured in mmHg
Heart rate | 2 hours after subarachnoid block
  number of heart beats per minute
APGAR score for assessment of the general state of the fetus | 10 minutes after delivery
  APGAR score of the fetus ranging from 0 to 10. the higher the value, the better he score
Incidence of reactive hypertension | 2 hours after spinal anesthesia
  Defined as the percentage of patients with increased systolic blood pressure more than 80% of the baseline reading
Umbilical arterial potential hydrogen (PH) | 10 minutes after delivery
  PH in the blood sample obtained from umbilical artery scaled from 1 to 14
Umbilical arterial Partial pressure of Carbon dioxide | 10 minutes after delivery
  in the blood sample obtained from umbilical artery measured in mmHg
incidence of nausea | 2 hours
  The percentage of patients with nausea
Incidence of vomiting | 2 hours
  The percentage of patients with nausea
Total phenylephrine consumption | 2 hours
  the total dose of phenylephrine consumed during the operation
Total norepinephrine consumption | 2 hours
  the total dose of norepinephrine consumed during the operation
Total ephedrine consumption | 2 hours
  the total dose of ephedrine consumed during the operation

CONTACTS AND LOCATIONS:
Overall Officials: Ahmed M Mukhtar, Professor, Study Director — Head of research committee section in anesthesia department
Locations (1):
- Cairo University, Cairo, Egypt

IPD SHARING:
Plan to Share IPD: No